CLINICAL TRIAL: NCT04224857
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single-Ascending Dose in Healthy Subjects and Multiple-Ascending Dose in Adult Patients With Ulcerative Colitis Study to Evaluate the Safety, Tolerability, PK and PD of Oral AMT-101
Brief Title: SAD/MAD Study in Healthy Subjects and Adults With UC to Evaluate Safety, Tolerability, PK, PD of AMT-101
Acronym: AURIGA1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Applied Molecular Transport (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMT-101-001
Record Dates: First submitted 2019-05-23; First posted 2020-01-13 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized to either receive AMT-101 or placebo
Who Masked: Participant, Investigator
Masking Description: matching placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AMT-101 (Experimental): AMT-101
  Interventions: Drug: AMT-101
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: AMT-101 — Single or daily dosing at doses A, B, C, D, E, F
  Other Names: no other name applicable
  Arms: AMT-101
Drug: Placebos — Single or daily dosing at doses A, B, C, D, E, F
  Other Names: no other name applicable
  Arms: Placebo

SUMMARY:
A randomized, double-blind placebo-controlled first in human study in approximately 36 male healthy subjects and approximately 20 male and female patients with active UC who have had an inadequate response to or demonstrated intolerance to 5-ASA.

DETAILED DESCRIPTION:
A randomized, double-blind placebo-controlled first in human study in approximately 36 male healthy subjects and approximately 20 male and female patients with active UC who have had an inadequate response to or demonstrated intolerance to 5-ASA.

Subjects may but are not required to have been exposed to corticosteroids, or immunosuppressive agents. In case the subject has been exposed to any of these treatments, he/she must have had either an inadequate response, failed response or demonstrated intolerance.

Patients may be

1. naïve to anti-TNFα therapy or
2. have failed or demonstrated intolerance to anti-TNF-α therapy.

ELIGIBILITY:
Inclusion Criteria:

PART A (Healthy Volunteers)

* Male subject in good health as determined by past medical history, physical examination, vital signs, ECG, and laboratory tests at screening
* Between 18 and 45 years of age, inclusive.
* Body Mass Index (BMI) between 18 and 30 kg/m2 (inclusive).

PART B (Adult Ulcerative Colitis)

* Male and Female patients 18 years and older
* Documented diagnosis of UC for at least 3 months duration
* Stable mild to moderate UC, as defined by the following criteria: Total Mayo score (excluding PGA) at least 3 but not greater than 7:
* Patients must have failed or demonstrated intolerance to aminosalicylates (e.g., 5-aminosalicylic acid, mesalamine)

Exclusion Criteria:

PART A and PART B

* Known hypersensitivity or allergy to AMT-101 or excipient contained in the drug formulation.
* Clinically significant abnormalities in laboratory test results (including complete blood count, chemistry panel including kidney panel, and urinalysis).

PART B

* Clinical findings of Crohn's disease
* A prior history of surgery for UC
* Prior use of integrin antagonists (vedolizumab, natalizumab), JAK kinase inhibitors (tofacitinib), cyclosporin or tacrolimus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Healthy Male Volunteers for Single Dose portion only
Enrollment: 52 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-emergent adverse events (safety and tolerability) | 14 days
  Single and multiple ascending doses of AMT-101 in healthy adult volunteers and patients with active UC by evaluation of incidence of treatment-related adverse events as assessed by CTCAE v4.03 and Modified Mayo Score criteria.

SECONDARY OUTCOMES:
Maximum plasma concentration (CMax) | 14 days
  To assess the pharmacokinetics of AMT-101 and Total IL-10 in healthy volunteers and subjects with UC.
Pharmacodynamics | 14 days
  To assess plasma IL-1Ra concentration in healthy volunteers and subjects with UC.

OTHER OUTCOMES:
Incidence of anti-drug antibodies against AMT-101 | 14 days
  Incidence of anti-drug antibodies against AMT-101 in healthy adult volunteers and subjects with UC.

CONTACTS AND LOCATIONS:
Overall Officials: Bittoo Kanwar, MD, Study Director — Applied Molecular Transport
Locations (4):
- LLC ARENSIA Exploratory Medicine, Tbilisi, Georgia
- Charité Research Organisation GmbH, Berlin, Germany
- ICS ARENSIA Exploratory Medicine SRL, Chisinau, Moldova
- Medical Center of Harmoniya krasy, Department of clinical trials, Kyiv, Ukraine